CLINICAL TRIAL: NCT05836311
Title: Single Perclose Escalation Technique for Vascular Closure in TAVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CLOSURE TAVI 1 VERSUS 2
Record Dates: First submitted 2023-04-13; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Aortic Valve Stenosis; Structural Valve Deterioration; Structural Valve Degeneration
Keywords: Residual Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with one Perclose Proglide: Patients undergoing transfemoral TAVI implantation treated with one Perclose Proglide Suture
  Interventions: Device: One Perclose Proglide Suture
- Patients treated with two Perclose Proglide Suture: Patients undergoing transfemoral TAVI implantation treated with two Perclose Proglide Suture
  Interventions: Device: Two Perclose Proglide Suture

INTERVENTIONS:
Device: One Perclose Proglide Suture — One Perclose Proglide Suture
  Groups: Patients treated with one Perclose Proglide
Device: Two Perclose Proglide Suture — One Perclose Proglide Suture
  Groups: Patients treated with two Perclose Proglide Suture

SUMMARY:
This study examines in the safety and efficacy of using a single Perclose escalation technique (SPET) using a single Perclose Proglide device to preclose and the need for a rescue device based on a control angiography at the end of the procedure, with a 6F femoral sheath.

DETAILED DESCRIPTION:
Percutaneous femoral access is the preferred access route for transcatheter aortic valve replacement (TAVR). The majority of experienced TAVR centers use two 6F Perclose ProGlide™ devices to close the primary vascular access site, deployed prior to upsizing sheath size with closure completed at the end of the case (the double "preclose" approach). A strategy of utilizing a single Perclose device to preclose may have advantages including fewer complications, complexity, and cost, but the safety of this is unknown. This study examines in the safety and efficacy of using a single Perclose escalation technique (SPET) using a single Perclose Proglide device to preclose and the need for a rescue device based on a control angiography at the end of the procedure, with a 6F femoral sheath. The use of Femoseal in mild bleedings, and a second Perclose Proglide for moderate to severe bleedings. Compare this SPET technique with double Preclose technique, with two historical cohorts of patients. One cohort of patients with SPET technique since started this technique, and a second cohort with double perclose technique prior to starting SPET technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients who have undergone Transfemoral TAVI implantation

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing transfemoral TAVI implantation in a single center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-19 (Estimated); Primary Completion 2025-02-19 (Estimated); Study Completion 2025-02-19 (Estimated)

PRIMARY OUTCOMES:
SAFETY:Incidence of Intrahospital Major Vascular Complications and Bleeding type 2 or type >2 (according to VARC 3 criteria) | 30 days
  Intrahospital Major Vascular Complications and Bleeding type 2 or type >2 (according to VARC 3 criteria)
EFFICACY:Incidence of successful femoral closure | 30 days
  Complete hemostasis at the puncture site with manual compression after the initial perclosure strategy

SECONDARY OUTCOMES:
Cost-effectiveness evaluation | 30 days
  Cost-effectiveness evaluation between two techniques
Incidence of vascular complications (according to VARC3 criteria) | 30 days
  Incidence of vascular complications (according to VARC3 criteria)
Incidence of bleeding (according to VARC3 criteria) | 30 days
  Incidence of bleeding (according to VARC3 criteria)
All-cause Mortality | 30 days
  All-cause Mortality 30 days after procedure
All-cause Mortality | 1 year
  All-cause Mortality 1 year after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall D'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodama A, Yamamoto M, Shimura T, Kagase A, Koyama Y, Tada N, Takagi K, Araki M, Yamanaka F, Shirai S, Watanabe Y, Hayashida K. Comparative data of single versus double proglide vascular preclose technique after percutaneous transfemoral transcatheter aortic valve implantation from the optimized catheter valvular intervention (OCEAN-TAVI) japanese multicenter registry. Catheter Cardiovasc Interv. 2017 Sep 1;90(3):E55-E62. doi: 10.1002/ccd.26686. Epub 2016 Oct 27. PMID 27785881
- [Background] Bazarbashi N, Ahuja K, Gad MM, Sammour YM, Kaur M, Karrthik A, Saad AM, Khubber S, Dhaliwal K, Mick SL, Navia JL, Puri R, Reed GW, Krishnaswamy A, Kapadia SR. The utilization of single versus double Perclose devices for transfemoral aortic valve replacement access site closure: Insights from Cleveland Clinic Aortic Valve Center. Catheter Cardiovasc Interv. 2020 Aug;96(2):442-447. doi: 10.1002/ccd.28585. Epub 2019 Nov 12. PMID 31713996